CLINICAL TRIAL: NCT07092449
Title: Pucotenlimab Combined With Chemotherapy (Nab-Paclitaxel + Tegafur + Carboplatin) in the Perioperative Treatment of Locally Advanced Gastroesophageal Junction Tumors, A Multi-center Prospective Study
Brief Title: Pucotenlimab Combined With Chemotherapy as Perioperative Treatment for Locally Advanced Gastroesophageal Junction Carcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT202505-06-KYB-05-XWK
Record Dates: First submitted 2025-07-08; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Gastroesophageal Junction; Gastric / Gastroesophageal Junction Adenocarcinoma; Neoadjuvant Chemoimmunotherapy; Adjuvant Therapy
Keywords: A Prospective Observational Study of Putilimab Combined with Chemotherapy in the Perioperative Treatment of Locally Advanced Gastroesophageal Junction Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group A (Experimental)
  Interventions: Drug: Neoadjuvant chemo-immunotherapy

INTERVENTIONS:
Drug: Neoadjuvant chemo-immunotherapy — Pucotenlimab combined with chemotherapy (Nab-Paclitaxel + Tegafur + Carboplatin)

SUMMARY:
This study is a prospective, multicenter, single-arm clinical trial.

The study intends to enroll patients with pathologically or cytologically confirmed resectable locally advanced gastroesophageal junction tumors (cT2N+M0 and cT3-4bNxM0) who have not received prior systemic therapy. After signing the informed consent and being screened to meet the inclusion and exclusion criteria, patients will receive 3 cycles of Pucotenlimab combined with chemotherapy (Nab-Paclitaxel + Tegafur + Carboplatin). Preoperative imaging evaluations will be performed 3 to 6 weeks after the final dose administration to assess the efficacy of neoadjuvant therapy and the feasibility of radical resection. Efficacy evaluation will be performed after radical surgery for locally advanced gastroesophageal junction tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent Provide written informed consent for the clinical study and biobank before any study-related procedures.
2. Age and Gender Male or female patients aged 18 to 75 years.
3. Disease Diagnosis Histologically confirmed resectable locally advanced gastroesophageal junction tumor.

   cTNM staging of cT2N+M0 or cT3-4bNxM0 based on endoscopic ultrasonography, contrast-enhanced CT/MRI (with endoscopic ultrasonography, diagnostic laparoscopy, or PET-CT as needed), corresponding to locally advanced gastroesophageal junction tumor per AJCC 9th edition, and deemed resectable by the investigator.
4. Prior Treatment History No prior systemic therapy for the current disease, including surgery, anti-tumor radiotherapy/chemotherapy, immunotherapy, etc.
5. Surgical Eligibility Agree to receive radical surgery and have no surgical contraindications as judged by surgeons.
6. Target Lesion Assessment At least one lesion (untreated with radiotherapy) meets RECIST 1.1 target lesion (TL) criteria.

   Tumor assessment must be performed via CT or MRI within 28 days before treatment.
7. Performance Status ECOG score of 0-1.
8. Life Expectancy Expected survival ≥ 3 months.
9. Organ Function Requirements

Laboratory parameters must meet the following within 14 days:

Absolute neutrophil count (ANC) ≥ 1.5×10⁹/L (without granulocyte colony-stimulating factor use).

Platelets ≥ 100×10⁹/L (without blood transfusion). Hemoglobin > 9 g/dL (without blood transfusion or erythropoietin use). Total bilirubin ≤ 1.5×ULN; if total bilirubin > 1.5×ULN, direct bilirubin must be ≤ ULN.

AST and ALT ≤ 2.5×ULN. Serum creatinine ≤ 1.5×ULN or creatinine clearance (Cockcroft-Gault formula) ≥ 60 mL/min.

Coagulation function: INR or PT ≤ 1.5×ULN. No severe thyroid dysfunction (as judged by the investigator). Cardiac function: NYHA class < 3; left ventricular ejection fraction ≥ 50%. 10. Contraceptive Measures and Pregnancy Testing

For female subjects of childbearing potential:

Negative urine or serum pregnancy test within 3 days before the first study drug administration (Cycle 1, Day 1). If urine test is inconclusive, a blood test is required.

Non-childbearing potential is defined as postmenopausal for ≥1 year, surgically sterilized, or having undergone hysterectomy.

All subjects (male and female) at risk of conception must use contraception with an annual failure rate < 1% throughout treatment and for 120 days after the last study drug administration (or 180 days after the last chemotherapy dose).

Exclusion Criteria:

1. Diagnosed with malignant diseases other than gastroesophageal junction tumors within 5 years before the first administration (excluding radically treated basal cell carcinoma of the skin, cutaneous squamous cell carcinoma, and/or carcinoma in situ after radical resection);
2. Known endoscopic evidence of active bleeding in the lesion;
3. Known evidence of distant metastasis;
4. Currently participating in therapeutic interventions of an interventional clinical study, or having received other drug therapies for malignant gastroesophageal junction tumors within 4 weeks before the first administration;
5. Having previously received the following therapies: anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs, or drugs targeting another stimulatory or co-inhibitory T-cell receptor (including but not limited to CTLA-4, OX-40, CD137, etc.), or chemotherapy (including but not limited to S-1);
6. Having received systemic treatment with Chinese patent medicines with anti-tumor indications or drugs with immunomodulatory effects (including thymosin, interferon, interleukin, excluding those used locally to control pleural effusion) within 2 weeks before the first administration;
7. Having had active autoimmune diseases requiring systemic treatment (such as disease-modifying drugs, glucocorticoids or immunosuppressants) within 2 years before the first administration. Alternative therapies (such as thyroxine, insulin, or physiological glucocorticoids for adrenal or pituitary insufficiency, etc.) are not considered systemic treatment;
8. Receiving systemic glucocorticoid therapy (excluding nasal spray, inhaled or other forms of topical glucocorticoids) or any other form of immunosuppressive therapy within 7 days before the first administration of the study; Note: The use of physiological doses of glucocorticoids (≤ 10 mg/day of prednisone or equivalent drugs) is allowed;
9. Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
10. Known history of allergy to putlizumab, chemotherapeutic drugs used in this study or their components;
11. Before starting treatment, not having fully recovered from toxicities and/or complications caused by any interventions (i.e., ≤ Grade 1 or returning to baseline, excluding fatigue or alopecia);
12. Known history of human immunodeficiency virus (HIV) infection (i.e., positive for HIV 1/2 antibodies);
13. Untreated active hepatitis B (defined as positive HBsAg with HBV-DNA copy number greater than the upper limit of normal of the laboratory in the research center);

Note: Hepatitis B subjects meeting the following criteria can also be enrolled:

1) HBV viral load < 1000 copies/ml (200 IU/ml) before the first administration, and subjects should receive anti-HBV treatment during the entire study period of chemotherapeutic drug treatment to avoid viral reactivation; 14. Subjects with active HCV infection (HCV antibody positive and HCV-RNA level above the lower limit of detection); 15. Having received a live vaccine within 30 days before the first administration (Cycle 1, Day 1); Note: Administration of inactivated viral vaccines for seasonal influenza within 30 days before the first administration is allowed; however, intranasal attenuated live influenza vaccines are not allowed; 16. Pregnant or lactating women; 17. Having any severe or uncontrollable systemic diseases, such as:

1. Significant and severely symptomatic abnormalities in resting electrocardiogram in terms of rhythm, conduction or morphology, such as complete left bundle branch block, second-degree or higher atrioventricular block, ventricular arrhythmias or atrial fibrillation;
2. Unstable angina pectoris, congestive heart failure, chronic heart failure with New York Heart Association (NYHA) class ≥ 2;
3. Any arterial thrombosis, embolism or ischemia occurring within 6 months before enrollment, such as myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack;
4. Poorly controlled hypertension with medication;
5. A history of non-infectious pneumonia requiring glucocorticoid treatment within 1 year before the first administration, or currently having clinically active interstitial lung disease;
6. Active pulmonary tuberculosis;
7. Having active or uncontrolled infections requiring systemic treatment;
8. Having clinically active diverticulitis, abdominal abscess, intestinal obstruction;
9. Liver diseases such as decompensated liver disease, acute or chronic active hepatitis;
10. Poorly controlled diabetes;
11. Patients with mental disorders who cannot cooperate with treatment; 18. Known dihydropyrimidine dehydrogenase deficiency; 19. Patients with gastrointestinal obstruction, or physiological dysfunction or malabsorption syndrome; Evidence of medical history, diseases, treatments or abnormal laboratory test values that may interfere with the study results, prevent the subjects from participating in the study throughout the process, or other situations that the researcher deems unsuitable for enrollment, or the researcher deems that there are other potential risks that make the subject unsuitable for participating in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
pCR | From enrollment to the end of treatment at 2 weeks
  Pathological complete response rate

SECONDARY OUTCOMES:
Major pathological response (MPR) Objective response rate (ORR) R0 resection rate Overall survival (OS) and 3-year overall survival rate (3-year OS) Disease-free survival (DFS) and 3-year disease-free survival rate (3-year DFS) Adverse events (AEs) | From enrollment to the end of treatment at 3 years
  Major pathological response (MPR) Objective response rate (ORR) R0 resection rate Overall survival (OS) and 3-year overall survival rate (3-year OS) Disease-free survival (DFS) and 3-year disease-free survival rate (3-year DFS) Adverse events (AEs)

OTHER OUTCOMES:
Objective response rate（ORR) | From enrollment to the end of treatment at 2 weeks
  The proportion of patients whose tumor volume shrinks to a predefined value and can maintain this minimum threshold for a required minimum duration is the sum of the proportions of complete response (CR) and partial response (PR). ORR = CR + PR
R0 resection rate | From enrollment to the end of treatment at 2 weeks
  Achievement of a curative resection rate of all surgery
overall survival | From enrollment to the end of treatment at 5 years
  The time from randomization to the patient's death from any cause
3-year OS | From enrollment to the end of treatment at 3 years
  Patients from randomization to the patient's death from any cause at 3 year rate in all patients
Progression-free Survival | From enrollment to the end of treatment at 5 years
  The time between the start of randomization and the occurrence of tumor progression (in any aspect) or death (due to any reason)
3-year PFS | From enrollment to the end of treatment at 3 years
  Patients from randomization to the patient's occurrence of tumor progressionrom any cause at 3 year rate in all patients
Adverse Event | From enrollment to the end of treatment at 5 years
  Adverse medical events experienced by subjects during the clinical trial process

IPD SHARING:
Plan to Share IPD: No